CLINICAL TRIAL: NCT01662388
Title: A Clinical Trial of Proximal Composite Restorations
Acronym: Automatrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Farhan Raza Khan, Assistant Professor, Dentistry, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 640-Sur-ERC-06; 640-Sur/ERC-06 (Other: Aga khan University)
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Class II Caries in Premolars
Keywords: proximal caries, composite restoration, proximal contact

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- automatrix band, Separation ring (Experimental): The prepared teeth received Automatrix band (similar to the control group, product code# 62422513). The Automatrix was burnished against the adjacent tooth gently. Anatomical wedges were applied in the proximal area and then the separation ring (BiTine® round ring by Palodent systems, Dentsply International, DE, USA product # 659040) placed with the help of retainer forceps.
  Interventions: Device: Separation ring; Device: automatrix band
- automatrix band (Active Comparator): Teeth received Automatrix band alone (Wide-Regular type, dimensions 7.9 mm height and 0.05mm thickness, product code # 62422513). It was secured on the prepared tooth and burnished against the adjacent tooth gently. Anatomical wedges were placed in the inter-proximal area gingival to the cavity preparation.
  Interventions: Device: automatrix band

INTERVENTIONS:
Device: Separation ring — Separation ring placed along with automatrix band
  Other Names: BiTine® Separation ring by Palodent, product # 659040)
  Arms: automatrix band, Separation ring
Device: automatrix band — band placed with a tightening device
  Other Names: circumferential automatrix band by Dentsply

SUMMARY:
Several techniques have been advocated to get good contacts in dental composite restorations including interdental separation ring. The investigators study focuses on using separation ring with circumferential matrix band instead of a sectional band. Moreover, the investigators have attempted to study proximal tightness and proximal contours of composite restoration as separate variables

DETAILED DESCRIPTION:
A total of 188 premolar teeth with proximal cavity to be assigned on alternate basis in two groups. Intervention group teeth received Automatrix band after cavity preparation followed by the separation ring using clamp while the control group received Automatrix band alone.

All teeth to be restored with P-60 composite restorative material(3M-ESPE Dental, USA). Outcome (proximal tightness) is determined by a blinded assessor just after the restoration.

ELIGIBILITY:
Inclusion Criteria:

* patients who had supra gingival Class II cavities in permanent premolars. Teeth with cavity isthmus less than one-third of intercuspal distance were inducted

Exclusion Criteria:

* Partially erupted teeth, teeth with non-carious tooth surface wear or with orthodontic bands or brackets or whose adjacent tooth continuous with the cavity side is missing were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
proximal tightness | 1 day (just after dental restoration)
  The tightness of the proximal contact area resulting from either of the two matrix band system. It was measured using a nine inch long nylon dental floss (Johnson and Johnson, USA).

SECONDARY OUTCOMES:
proximal contours | 1 day (just after restoration placement)
  To be examined clinically with an explorer and mouth mirror and then on the periapical radiograph by the blinded co investigator.

OTHER OUTCOMES:
Overhang of the restoration | 1 day (just after the restoration placement)
  To be examined clinically with an explorer and mouth mirror and then on the periapical radiograph by the blinded co investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Farhan R Khan, FCPS, Principal Investigator — AKU
Locations (1):
- Dental Clinics, Aga Khan University Hospital, Karachi, Sindh, Pakistan